CLINICAL TRIAL: NCT00259753
Title: A Phase II, Randomized, Double-Masked, Controlled, Dose Comparison Study of Cand5 for Intravitreal Injection for the Treatment of Subfoveal Choroidal Neovascularization Associated With Wet Age-Related Macular Degeneration
Brief Title: Safety and Efficacy Study of Small Interfering Ribonucleic Acid (RNA) Molecule (Cand5) to Treat Wet Age-Related Macular Degeneration
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OPKO Health, Inc. (Industry)
Responsible Party: Denis O'Shaughnessy, Opko Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACU201
Record Dates: First submitted 2005-11-30; First posted 2005-12-01 (Estimated); Last update posted 2008-08-05 (Estimated); Status verified 2008-07

CONDITIONS: Macular Degeneration
Keywords: Wet Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — bevasiranib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): 0.2 mg/eye
  Interventions: Drug: Bevasiranib
- 2 (Experimental): 1.5 mg/eye
  Interventions: Drug: Bevasiranib
- 3 (Experimental): 3.0 mg/eye
  Interventions: Drug: Bevasiranib

INTERVENTIONS:
Drug: Bevasiranib
  Other Names: Cand5

SUMMARY:
The objective of this study is to evaluate the safety and preliminary efficacy of three doses of Cand5. Cand5, a small interfering RNA molecule that selectively silences the mRNA encoding for VEGF.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have subfoveal classic, predominantly classic, or minimally classic lesions, secondary to AMD.
2. Patients must have ETDRS best corrected visual acuity of 64 to 24 letters (20/50 to 20/320 Snellen Equivalent) in the study eye.
3. Patients must be age 50 or older

Exclusion Criteria:

1. Patients who have received prior treatment with any investigational new drug or device for wet AMD in the study eye within 24 weeks of the screening visit.
2. Patients with advanced glaucoma (greater than 0.8 cup:disk) or intraocular pressure above 22 mmHg in the study eye.
3. Patients with any retinal vasculopathies, including diabetic retinopathy, retinal vein occlusions, etc. in the study eye.
4. Patients with any subfoveal scarring, atrophy, or hemorrhage in the study eye.
5. Patients whose CNV lesion in the study eye contains more than 25% scarring and/or atrophy.
6. Patients who have undergone any extrafoveal/juxtafoveal laser treatment of the study eye within two weeks prior to the screening visit.
7. Patients who received treatment with an investigational drug within 4 weeks prior to the screening visit.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2005-07; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
change from baseline at the 12-week evaluation in macular edema as measured by optical coherence tomography. | 12 week

SECONDARY OUTCOMES:
The secondary endpoint is the mean BCVA line/letters change from baseline at the 12-week evaluation. | 12 week

CONTACTS AND LOCATIONS:
Overall Officials: Denis O'Shaughnessy, PHD, Study Director — Opko Health
Locations (23):
- United States (23):
  - Acuity Participating Site, Phoenix, Arizona
  - Retina Centers PC, Tucson, Arizona
  - Sall Research Medical Center, Artesia, California
  - Bay Area Retina Associates, Walnut Creek, California
  - Florida Eye Microsurgical Institute, Inc., Boynton Beach, Florida
  - Retina Specialist, Towson, Maryland
  - Vitreo-Retinal Associates PC, Grand Rapids, Michigan
  - Associated Retinal Consultants, Grand Rapids, Michigan
  - Associated Retinal Consultants, P.C., Royal Oak, Michigan
  - VitreoRetinal Surgery, P.A., Edina, Minnesota
  - Eye Foundation of Kansas City, UMKC School of Medicine, Kansas City, Missouri
  - Retina-Vitreous Center, Lakewood, New Jersey
  - Retina-Vitreous Consultants, Livingston, New Jersey
  - OCLI, Lynbrook, New York
  - LuEsther T. Mertz Retinal Research Center, New York, New York
  - Southeast Clinical Research, Charlotte, North Carolina
  - Retina Associates of Cleveland, Beachwood, Ohio
  - Retina Associates of Cleveland, Inc., Lakewood, Ohio
  - Black Hills Eye Institute, Rapid City, South Dakota
  - Retina Reseach Center, Austin, Texas
  - Ophthalmology Associates, Fort Worth, Texas
  - Vitreoretinal Consultants Houston TX, Houston, Texas
  - Medical College of Wisconsin Eye Institute, Milwaukee, Wisconsin

REFERENCES:
- See also: Sponsor — http://www.opko.com